CLINICAL TRIAL: NCT05389644
Title: Circuit-specific Neuromodulation for the Treatment of Apathy in Alzheimer's Disease
Brief Title: TMS as a Treatment for Apathy in Alzheimer's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to fulfill recruitment goals
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mark C. Eldaief, MD, Assistant Professor of Neurology, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022P001058
Record Dates: First submitted 2022-04-19; First posted 2022-05-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease; Apathy in Dementia
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This study will involve a within-subject crossover design. Every subject will undergo three interventions.
Who Masked: Participant
Masking Description: Participants will receive active stimulation to two sites as well as sham stimulation to a third site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dorsal circuit (DLPFC) stimulation (Experimental): This arm will involve stimulation of the dorsal apathy-relevant circuit. Specifically, a target will be individually selected based on resting-state functional connectivity with a given subject's dorsal striatum.
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- Ventral circuit (vmPFC) stimulation (Experimental): This arm will involve stimulation of the ventral apathy-relevant circuit. Specifically, a target will be individually selected based on resting-state functional connectivity with a given subject's ventral striatum.
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- Sham stimulation (Sham Comparator): This arm will involve sham stimulation to a prefrontal target.
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation (iTBS) — iTBS is a form of repetitive TMS. TMS is a form of non-invasive brain stimulation. In this modality, a current is rapidly passed through a TMS coil. This coil is placed on a subject's scalp. The rapidly discharging current creates a magnetic field perpendicular to the plane of the coil. This magnetic field diffuses through the subject's scalp and skull until it reaches the brain parenchyma. There, it causes focal neuronal depolarization.
  Other Names: Transcranial Magnetic Stimulation (TMS)

SUMMARY:
This proposal will demonstrate that non-invasive brain stimulation is able to modulate cortico-striatal circuits in neurodegenerative patients with apathy, and that doing so results in circuit-specific increases in FC and DA availability. These circuit changes will be accompanied by changes in specific behavioral dimensions of apathy. This work will lead to larger studies which develop personalized, circuit-specific neuromodulation strategies for AD patients suffering from this intractable neuropsychiatric symptom.

DETAILED DESCRIPTION:
Apathy is among the most common neuropsychiatric symptoms in Alzheimer's Disease (AD), with prevalence estimates up to 72%. Apathy in AD is associated with significant morbidity, high caregiver burden, and is correlated with disease severity. While other behavioral symptoms are clinically addressable in AD, there are currently no effective treatments for apathy.

Executive aspects of apathy involve deficits in goal-directed planning, rule maintenance, cognitive flexibility, and set-shifting. Motivational aspects of apathy involve reward anticipation, valuation of the effort needed to achieve a goal, and the consummatory experience once a goal is achieved. Importantly, these discrete cognitive-behavioral dimensions can be mapped onto discrete fronto-striatal circuits. For example, executive deficits are likely to map onto dorsolateral prefrontal-striatal loops (a dorsal apathy-related circuit). In contrast, motivational processing is localizable to projections between the ventral striatum (VS) and the anterior cingulate cortex (ACC), ventromedial prefrontal cortex (vmPFC) and orbitofrontal cortex (OFC) (a ventral apathy-related circuit).

Dopamine (DA) supports processing in both the dorsal and ventral circuits, and there is voluminous evidence that DA plays roles in encoding reward prediction/valuation and motivation. For example, the ventral circuit receives dense monosynaptic dopaminergic projections from the ventral tegmental area, and several studies have invoked this pathway in reward processing. DA also plays a role in executive function. Moreover, apathy is observed in patients with disorders of DA availability, in patients taking DA antagonists and with lesions in the meso-cortico-limbic pathway. More specifically, AD patients exhibit decreased striatal DA availability. Taken together, decreased DA transmission in the dorsal and ventral circuits represent putative neurochemical mechanisms for apathy in AD.

Repetitive transcranial magnetic stimulation (rTMS) is capable of modulating fMRI resting-state functional connectivity (FC) in a circuit-specific manner. For example, our group, as well as others, have demonstrated the feasibility of modulating network FC through stimulation of a cortically accessible network node. Other studies have demonstrated behavioral changes with circuit-specific neuromodulation. Prefrontal rTMS can also modulate monoaminergic neurotransmitter release in a regionally specific way. For example, intermittent theta burst stimulation (iTBS, a form of rTMS) increases tonic endogenous DA release in animal models, and this effect can be blocked by DA receptor antagonists. There is also evidence in humans that topographically specific changes in DA release can be elicited based on the circuit stimulated. For instance, Strafella and colleagues used an rTMS-11C- raclopride paradigm to show regionally specific changes in DA availability following dorsolateral prefrontal (dlPFC) stimulation and primary motor cortex stimulation, respectively. We recently extended this work by employing a combined MRI-PET paradigm with 11C-raclopride. In that protocol, three subjects underwent iTBS to two adjacent dlPFC targets. These targets were functionally identified by the maximal FC with two dorsal striatal regions: the left caudate and left putamen, and these were seeded based on coordinates derived from large datasets. Targets were stimulated based on modeled E- field distributions. As predicted, iTBS induced regionally specific changes in striatal DA availability, with changes in 11C- raclopride binding potentials (BPND) occurring at the sites of maximal FC with the respective iTBS targets.

Aim 1: To optimize rTMS targeting of apathy-relevant circuits in AD patients with apathy: Hypothesis 1.1: FC estimates, acquired with accelerated multi-band imaging, will identify, on an individualized basis, rTMS accessible cortical targets (e.g., in vmPFC/mOFC and in dlPFC) which are most functionally coupled to relevant striatal regions (e.g., the VS and dorsal caudate) in a group of AD patients with apathy. Hypothesis 1.2: State-of-the-art E-field modeling will optimize coil position and orientation needed to best stimulate the apathy-relevant circuits. Modeling will be informed by (a) structural estimates of cortical atrophy, (b) diffusion MRI tractography estimates of white matter fiber bundles from cortical targets.

Aim 2: To use rTMS to differentially modulate FC in apathy-relevant circuits in AD patients with apathy: Hypothesis 2.1: rTMS to the dorsal circuit will increase FC specifically in the dorsal circuit. Hypothesis 2.2: rTMS to the ventral circuit will increase FC specifically in the ventral circuit. Hypothesis 2.3: Sham rTMS will not affect FC in either circuit.

Aim 3: To use rTMS to differentially modulate DA in apathy-relevant circuits in AD patients with apathy: Hypothesis 3.1: rTMS to the dorsal circuit will increase DA availability, (as measured by changes in 11C- raclopride binding potential (BPND)), specifically in the dorsal circuit. Hypothesis 3.2: rTMS to the ventral circuit will increase DA availability specifically in the ventral circuit. Hypothesis 3.3: Sham rTMS will not affect DA availability in either circuit.

Aim 4: To assess behavioral changes induced by modulation of apathy-relevant circuits in AD patients: Hypothesis 4.1: rTMS to the dorsal circuit will selectively improve executive measures of goal-directed behavior, as assessed by fMRI task performance on planning portions of the PACT. Hypothesis 4.2: rTMS to the vental circuit will selectively improve motivation and reward anticipation, as assessed by fMRI task performance and activation on motivational parts of the PACT, and on mood scales. Hypothesis 4.3: Sham rTMS will have no impact on fMRI task performance or activation, nor on mood scales.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80.
2. A clinical diagnosis of Alzheimer's disease, including atypical variants of this (e.g., the behavioral/dysexecutive variant, the logopenic Primary Progressive Aphasia variant, Posterior Cortical Atrophy variant, etc.).
3. Clinical Dementia Rating of 0.5 or mild 1.0 (MMSE equal to or greater than 22).
4. Patients must be accompanied to visits by a study partner/informant (usually a spouse or adult child).
5. Prominent symptoms of apathy reported by their primary caregiver/informant and verified with a score of greater than or equal to 45 on the informant version of the Apathy Evaluation Scale (AES-I).

Exclusion Criteria:

1. Any contraindication to MR-PET scanning (e.g., pacemakers, implanted metal, aneurysm clips, etc.)
2. Any contraindication to receiving TMS (e.g., a history of seizures, cochlear implants)
3. Involvement in any PET studies within 12 months.
4. Clinical dependence on psychotropic medications believed to affect dopamine binding (e.g., certain antidepressants or especially neuroleptics). If the patient is clinically able to temporarily wean off of these, they will be included after the medication has been discontinued and fully eliminated (e.g., a duration of five half-lives). Subjects will also be excluded if they have a history of long-term use of these agents (particularly neuroleptics).
5. Concurrent use of tobacco or illicit drugs, particularly those affecting dopamine transmission. Patients will be asked to refrain from using caffeine the morning of experimental procedures.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Changes in resting-state connectivity (FC). | 1 hour
  Changes in circuit-specific FC will be assessed with functional magnetic resonance imaging (fMRI) before and after iTBS.
Changes in dopamine (DA) availability. | 1 hour
  Changes in DA availability after iTBS to each target will be measured by changes in 11C- raclopride binding potential (BPND)
Changes in fMRI activation on an apathy related task | 1 hour
  Changes in fMRI blood oxygenation level dependent activation on the Philadelphia Apathy Computerized Test (PACT)
Changes in performance on an apathy related task | 1 hour
  Changes in reaction times on the Philadelphia Apathy Computerized Test (PACT)
Changes in scores on an apathy scale | 1 hour
  Changes in scores on the Apathy Evaluation Scale (AES); range 0-36, higher scores indicating more apathy.
Changes in mood scores | 1 hour
  Changes in scores on the Profile of Mood States (POMS); range 0-20, higher scores indicating less apathy.
Changes in mood scores | 1 hour
  Changes in scores on the Positive and Negative Affect Scale (PANAS); range 10-50, higher scores indicating less apathy.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Eldaief, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Martinos Center for Biomedical Imaging/Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No